CLINICAL TRIAL: NCT02664467
Title: Chronobiology, Sleep Related Risk Factors and Light Therapy in Perinatal Depression: the Life-ON Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Regionale di Lugano (Other)
Collaborators: University of Bologna (Other); University of Milan (Other); University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Mauro Manconi, Dr. med. Mauro Manconi, Ospedale Regionale di Lugano
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ORLugano
Record Dates: First submitted 2016-01-13; First posted 2016-01-27 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Depression; Depression, Postpartum; Depressive Disorder; Depressive Disorder, Major; Mood Disorders; Pregnancy Complications; Puerperal Disorders
MeSH Terms: conditions — Depression; Depression, Postpartum; Depressive Disorder; Depressive Disorder, Major; Mood Disorders; Pregnancy Complications; Puerperal Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bright light therapy (BLT) (Experimental): Bright light therapy (10'000 lux) for 30 minutes after wake-up using Philips EnergyUp EnergyLight HF3419/01
  Interventions: Device: Philips EnergyUp EnergyLight HF3419/01
- Placebo dim light (Placebo Comparator): Placebo dim light (50 lux) for 30 minutes after wake-up using Philips EnergyUp EnergyLight HF3419/01
  Interventions: Device: Philips EnergyUp EnergyLight HF3419/01

INTERVENTIONS:
Device: Philips EnergyUp EnergyLight HF3419/01 — Bright light therapy (10'000 lux) for 60 minutes after wake-up
  Arms: Bright light therapy (BLT)
Device: Philips EnergyUp EnergyLight HF3419/01 — Placebo dim light (500 lux) for 60 minutes after wake-up
  Arms: Placebo dim light

SUMMARY:
In a 3 years longitudinal, observational, multicentre study, about 500 women will be recruited and followed-up from early pregnancy (10-15 gestational week) until 12 months after delivery. The primary aim of the present study is to systematically explore and characterize risk factors for perinatal depression (PND) by prospective sleep assessment (using wrist actigraphy, polysomnography and various sleep questionnaires) and blood based analysis of potential markers during the perinatal period (Life-ON study). Secondary aims are to explore the relationship between specific genetic polymorphisms and PND (substudy Life-ON1), to investigate the effectiveness of BLT in treating PND (substudy Life-ON2) and to test whether a short term trial of BLT during pregnancy can prevent PND (substudy Life-ON3).

The characterization of specific predictive and risk factors for PND may substantially contribute to improve preventive medical and social strategies for the affected women. The study results are expected to promote a better understanding of the relationship between sleep disorders and the development of PND and to confirm, in a large sample of women, the safety and efficacy of BLT both in prevention and treatment of PND.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy
* Normal ocular function
* Gestational age between 10 to 15 weeks at time of screening
* Written informed consent

Exclusion Criteria:

* Diagnosis of bipolar I or II disorder (DSM-5)
* Recent history (less than 6 months) or current major depression or an Edinburgh Postnatal Depression Scale (EPDS) score > 12 at time of inclusion
* Any psychotic episode, substance abuse, recent history of suicide attempt (less than 12 months)
* Use of antidepressants or other pharmacologic treatments for depression in the last 6 months
* Fetal malformations and intrauterine fetal death

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Change in Depression Score as assessed by the Edinburgh Postnatal Depression Scale (EPDS) | during 6 weeks of light treatment plus 12 months observation
Change in Depression Score as assessed by the Hamilton Depression Rating scale - 21 items (HDRS-21) | during 6 weeks of light treatment plus 12 months observation
Change in Depression Score as assessed by the Montgomery-Asberg Depression Rating Scale (MADRS) | during 6 weeks of light treatment plus 12 months observation

SECONDARY OUTCOMES:
Objective sleep-related markers and risk factors for perinatal depression as assessed by home polysomnography | at 23th-25th week of gestation
Objective sleep-related markers and risk factors for perinatal depression as assessed by wrist actigraphy | observation over a period of 2 years
Analysis of genetic risk factors for perinatal depression by single blood test | at 23th-25th week of gestation
Subjective mood changes as assessed by the Visual Analog Scale for Depression (VAS) | during 6 weeks of light treatment plus 12 months observation
Number of participants with treatment-related adverse events as assessed by the Systematic Assessment for Treatment Emergent Events (SAFTEE) | during 6 weeks of light treatment plus 12 months observation

CONTACTS AND LOCATIONS:
Locations (1):
- Neurocenter of Southern Switzerland, Lugano, Canton Ticino, Switzerland

REFERENCES:
- [Derived] Garbazza C, Cirignotta F, D'Agostino A, Cicolin A, Hackethal S, Wirz-Justice A, Cajochen C, Manconi M; "Life-ON" study group. Sustained remission from perinatal depression after bright light therapy: A pilot randomised, placebo-controlled trial. Acta Psychiatr Scand. 2022 Oct;146(4):350-356. doi: 10.1111/acps.13482. Epub 2022 Aug 3. PMID 35876837
- [Derived] Baiardi S, Cirignotta F, Cicolin A, Garbazza C, D'Agostino A, Gambini O, Giordano A, Canevini M, Zambrelli E, Marconi AM, Mondini S, Borgwardt S, Cajochen C, Rizzo N, Manconi M. Chronobiology, sleep-related risk factors and light therapy in perinatal depression: the "Life-ON" project. BMC Psychiatry. 2016 Nov 4;16(1):374. doi: 10.1186/s12888-016-1086-0. PMID 27814712